CLINICAL TRIAL: NCT00851929
Title: Ambrisentan (Letairis) for Sarcoidosis Associated Pulmonary Hypertension
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Marc A. Judson, M.D., Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17747
Record Dates: First submitted 2009-02-24; First posted 2009-02-26 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Sarcoidosis; Pulmonary Hypertension
Keywords: sarcoidosis; pulmonary hypertension; dyspnea; sarcoidosis associated pulmonary hypertension
MeSH Terms: conditions — Sarcoidosis; Hypertension, Pulmonary; Dyspnea | interventions — ambrisentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sarcoidosis associated pulmonary hypertension (Experimental): sarcoidosis associated pulmonary hypertension
  Interventions: Drug: Ambrisentan

INTERVENTIONS:
Drug: Ambrisentan — ambrisentan 5 mg/day for month month, then 10 mg/day for 3 additional months
  Other Names: Letairis

SUMMARY:
Hypothesis: Ambrisentan (Letairis ®) is safe and effective in treating pulmonary hypertension in patients with Sarcoidosis

DETAILED DESCRIPTION:
Primary Endpoint: Change in 6 minute walk distance.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven sarcoidosis
* Mean pulmonary artery pressure > 25 mmHg at rest and greater than 30 mmHg with exercise by right heart catheterization within 1 year prior to entry into study
* Pulmonary capillary wedge pressure ≤ 15 mmHg
* PVR values >3.0 Woods units
* Forced vital capacity (FVC) >40%
* WHO functional class II or III
* Stable sarcoidosis treatment regimen for three months prior to entry into study
* 6 minute walk distance between 150-450 meters
* Stable dose of antihypertensive medications
* On no other medication to treat PAH (sildenafil, tadalafil, vardenafil, treprostinil, epoprostenol, iloprost, bosentan, sitaxsentan) within one month prior to enrollment and during duration of the study
* Non-pregnant females

Exclusion Criteria:

* Exercise limitation related to a non-cardiopulmonary reason (e.g. arthritis)
* Severe systemic hypertension > 170/95
* Patients with congestive heart failure (left ventricular dysfunction) or primary right ventricular dysfunction
* Anticipation by the investigator for escalation in sarcoidosis treatment during the course of the study
* Pulmonary hypertension related to etiology other than sarcoidosis (i.e. HIV, scleroderma, etc.)
* Use within 1 month of an endothelin receptor antagonists (bosentan, sitaxsentan).
* WHO functional class IV status
* Patients with significant left ventricular dysfunction
* Significant liver dysfunction not due to sarcoidosis.
* Patients with severe other organ disease felt by investigators to impact on survival during the course of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-11; Primary Completion 2011-04 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change in 6 minute walk distance. | 4 months of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Judson, MD, Principal Investigator — Medical University of South Carolina; Don C Rockey, MD, Study Chair — Medical University of South Carolina
Locations (2):
- United States (2):
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Medical Univerrsity of South Carolina, Charleston, South Carolina